CLINICAL TRIAL: NCT02461888
Title: A Randomised Phase II Trial of Cyclophosphamide and Dexamethasone in Combination With Ixazomib in Relapsed or Refractory Multiple Myeloma (RRMM) Patients Who Have Relapsed After Treatment With Thalidomide, Lenalidomide and Bortezomib.
Brief Title: Phase II Randomised Trial of Cyclophosphamide & Dexamethasone in Combination With Ixazomib in Relapsed or Refractory Multiple Myeloma.
Acronym: MUKEight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Myeloma UK (Other); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Gordon Cook, Chief Investigator, University of Leeds
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM13/10993
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Refractory; Cyclophosphamide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — ixazomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ixazomib, CD (Experimental): Ixazomib, cyclophosphamide and dexamethasone (ICD) will be administered as part of a 28 days cycle until disease progression, intolerance, toxicity or withdrawal.
  Dosing schedule:
  * Ixazomib 4mg orally on days 1, 8 and 15
  * Cyclophosphamide 500mg orally on days 1, 8 and 15
  * Dexamethasone 40mg orally on days 1-4 and 12-15
  Interventions: Drug: Ixazomib; Drug: Cyclophosphamide; Drug: Dexamethasone
- CD (Active Comparator): Cyclophosphamide and dexamethasone (CD) will be administered as part of a 28 days cycle until disease progression, intolerance, toxicity or withdrawal.
  Dosing schedule:
  * Cyclophosphamide 500mg orally on days 1, 8 and 15
  * Dexamethasone 40mg orally on days 1-4 and 12-15
  Interventions: Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Chemotherapy
  Arms: Ixazomib, CD
Drug: Cyclophosphamide — Chemotherapy
Drug: Dexamethasone — Chemotherapy

SUMMARY:
This study evaluates a new treatment combination of ixazomib with cyclophosphamide and dexamethasone in relapsed or refractory multiple myeloma. Participants will either receive ixazomib with cyclophosphamide and dexamethasone or cyclophosphamide and dexamethasone alone.

DETAILED DESCRIPTION:
Cyclophosphamide and dexamethasone are very commonly used in the treatment of multiple myeloma and are often given with a third drug (e.g. thalidomide, lenalidomide or bortezomib). The combination of conventional and new drugs has provided benefits in both overall survival and progression free survival, however there are few treatments available for patients who have not responded well (refractory) to their previous treatment or who need further treatment because their myeloma has come back (relapsed). Thus there is a need for new agents for these patients.

The development of ixazomib provides the opportunity to increase anti-tumour activity against a wider range of tumour types. Early clinical trials data suggests it has anti-tumour activity in heavily pre-treated multiple myeloma patients with durable responses/disease control and is generally well tolerated.

Cyclophosphamide and dexamethasone are both predominantly used in treatment of multiple myeloma and for patients with relapsed or refractory multiple myelomas (RRMM), who have relapsed after bortezomib and lenalidomide. Therefore the evaluation of ixazomib in combination with cyclophosphamide and dexamethasone is the most valuable and practical option for patients.

The primary end point of this study is progression-free survival (PFS). Secondary end points include toxicity and safety.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent and willing to follow study protocol assessments
* Aged 18 years or over
* Participants with confirmed multiple myeloma based on International Myeloma Working Group (IMWG) criteria, 2009
* Measurable disease
* Participants with relapsed or relapsed refractory myeloma and now require further treatment following exposure to thalidomide, lenalidomide and bortezomib regardless of response to these
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Required laboratory values within 14 days prior to Randomisation:
* Platelet count ≥50x109/L. Platelet support is permitted within 14 days prior to Randomisation
* Absolute neutrophil count ≥1.0 x 109/L
* Haemoglobin > 9 g/dL. Blood support is permitted
* Alanine aminotransferase (ALT) and / or Aspartate aminotransferase (AST) ≤3 x upper limit of normal
* Creatinine clearance ≥ 30 ml/min (using Cockcroft Gault formula)
* Bilirubin ≤1.5 x upper limit of normal
* Both non-sterilised and sterilised females and males of reproductive age should use effective methods of contraception during the entire trial treatment (including treatment breaks) and up to 90 days after the last dose of trial treatment
* Post allograft patients may be included

Exclusion Criteria:

* Those with non-measurable disease
* Those with a solitary bone or solitary extramedullary plasmacytoma
* Plasma cell leukaemia
* Prior malignancy other than those treated with curative surgery.
* Participants with a known or underlying uncontrolled concurrent illness that, in the investigators opinion, would make the administration of the study drug hazardous or circumstances that could limit compliance with the study
* Patients who have previously received MLN9708/Ixazomib in a trial. Previous experimental agents or approved anti-tumour treatment within 30 days before the date of randomisation.
* A maximum of 160mg of dexamethasone (in 40mg blocks) may be given between screening and the beginning of treatment if medically required but should be stopped before trial treatment starts. Bisphosphonates for bone disease and radiotherapy for palliative intent are also permitted
* Participants with a history of a refractory nausea, diarrhoea, vomiting, malabsorption, gastrointestinal surgery or other procedures that might, in the opinion of the Investigator, interfere with the absorption or swallowing of the study drug(s)
* Peripheral neuropathy of ≥ grade 2 severity
* Gastrointestinal disorders that may interfere with absorption of the study drug
* Active symptomatic fungal, bacterial, and/or viral infection including known active HIV or known viral (A, B or C) hepatitis
* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Systemic treatment, within 14 days before the first dose of MLN9708, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Major surgery within 14 days prior to the date of randomisation
* Radiotherapy within 14 days prior to randomisation
* Disease involving the Central Nervous System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2025-01-19 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From randomisation to first documented evidence of disease progression or death, up to 36 months.

SECONDARY OUTCOMES:
Response to treatment | From initial trial treatment until at least partial response is achieved, up to 36 months..
Maximum response | From initial trial treatment each of the response categories are achieved stringent complete response, complete response, very good partial response, partial response, minimal response or stable disease, up to 36 months.
Time to progression | From randomisation to first documented evidence of disease progression, up to 36 months..
Time to maximum response | From randomisation until the participant achieves any of the categories stringent complete response, complete response, very good partial response, partial response, minimal response or stable disease, up to 36 months.
Response duration | From the first observation of at least partial response until disease progression, up to 36 months.
Overall survival | From randomisation to death, up to 36 months.
Evaluate the safety and toxicity as measured by adverse reactions and serious adverse event reporting. | From consent until 28 days after the last dose of trial treatment, up to 36 months.
Treatment compliance measured by treatment delays and missed treatment doses. | From initial treatment received as per protocol until withdrawal from treatment, up to 36 months.
Quality of life measured by the completion of EQ-5D and EORTC QLQ-C30 questionnaires | Completed every 3 months from consent until disease progression, up to 36 months.
Cost effectiveness of treatment assessed by health economic evaluations. | From consent up to 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Cook, Principal Investigator — Leeds Teaching Hospitals NHS Trust
Locations (18):
- United Kingdom (18):
  - Queen Elizabeth Medical Centre, Birmingham
  - Heart of England NHS Foundation Trust, Birmingham
  - Royal Bournemouth General Hospital, Bournemouth
  - University Hospital Bristol NHS Foundation Trust, Bristol
  - North Tees and Hartlepool NHS Foundation Trust, Hartlepool
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Liverpool and Broadgreen University Hospital NHS Trust, Liverpool
  - Barts and the London NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's and St Thomas's NHS Foundation Trust, London
  - Royal Marsden Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospital NHS Trust, Nottingham
  - Churchill Hospital, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Southampton University Hospital NHS Trust, Southampton
  - The Royal Wolverhampton Hospital NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided